CLINICAL TRIAL: NCT06897254
Title: Outcomes of Acute Kidney Injury Requiring Renal Replacement Therapy in a Tertiary Level Teaching Hospital in Nepal: a Registry Based Retrospective Study
Brief Title: Outcomes of Critically Ill Patients Undergoing RRT- a Registry Based Study.
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Bipin Karki, Primary investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 518(6-11)E2-079/080
Record Dates: First submitted 2025-03-16; First posted 2025-03-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Renal Replacement Therapies; Outcome Assessment
Keywords: renal replacement therapy; hemodialysis; intensive care unit; outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RRT: Patients undergoing renal replacement therapy
- NRRT: Patients not undergoing renal replacement therapy

SUMMARY:
Rationale: Acute kidney injury (AKI) requiring renal replacement therapy (RRT) is a frequently occurring entity among critically ill patients. This study aims to determine the outcomes of patients undergoing renal replacement therapy in the ICU.

Study Objective: To find the outcomes of patients undergoing RRT in the ICU in terms of mortality and length of ICU stay.

Design: A registry based, retrospective, descriptive study. Sample size: Convenience sampling of all the patients who require RRT during the ICU stay.

Duration: Retrospective data from three years January 1, 2020 to December 30, 2023.

Place: Intensive care units (ICUs) of the Department of Critical Care Medicine, Tribhuvan University Teaching Hospital (TUTH).

Interventions: Not applicable Expected results: The study will help determine the outcomes of the critically ill patients undergoing RRT in a low middle income country ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Admission to the ICU
* All patients undergoing RRT during ICU stay

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU requiring renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ICU mortality | A the end of 3 years

SECONDARY OUTCOMES:
Treatment limitations | At the end of 3 years
  Patients who receiving treatment limitation orders (Leave against medical advice, do not resuscitate/do not intubate, withdrawal of treatment orders)

OTHER OUTCOMES:
LOS-ICU | At the end of 3 years
  Number of days admitted to the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Mahārājgañj, Bagmati, Nepal

REFERENCES:
- [Background] Cerda J, Mohan S, Garcia-Garcia G, Jha V, Samavedam S, Gowrishankar S, Bagga A, Chakravarthi R, Mehta R. Acute Kidney Injury Recognition in Low- and Middle-Income Countries. Kidney Int Rep. 2017 Jul;2(4):530-543. doi: 10.1016/j.ekir.2017.04.009. Epub 2017 Apr 25. PMID 29034358
- [Background] Andonovic M, Traynor JP, Shaw M, Sim MAB, Mark PB, Puxty KA. Short- and long-term outcomes of intensive care patients with acute kidney disease. EClinicalMedicine. 2022 Feb 12;44:101291. doi: 10.1016/j.eclinm.2022.101291. eCollection 2022 Feb. PMID 35198917